CLINICAL TRIAL: NCT03415568
Title: The Effects of Functional Edible Oil (MCDG) on Reducing Body Fat of Overweight or Obesity Subjects (Part.2)
Brief Title: Effects of MCDG Oil on Postprandial Lipid Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Jong Ho Lee, Professor, Yonsei University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DOP_OFTT
Record Dates: First submitted 2018-01-15; First posted 2018-01-30 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hyperlipidemias; Triglycerides High
Keywords: Postprandial lipid metabolism; Medium-chain triglycerides; Diacylglycerols; Serum triglycerides; Chylomicron triglycerides
MeSH Terms: conditions — Hyperlipidemias; Hypertriglyceridemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCT consumption (Placebo Comparator): Muffin that contains 15g of long-chain triglyceride (LCT) oils were provided to conduct 6-h meal tolerance test.
  Interventions: Dietary Supplement: LCT oil
- MCDG consumption (Experimental): Muffin that contains 15g of the mixture of medium-chain triglyceride and diacylglycerol (MCDG) oils were provided to conduct 6-h meal tolerance test.
  Interventions: Dietary Supplement: MCDG oil

INTERVENTIONS:
Dietary Supplement: LCT oil — LCT muffin was provided to the study participants. The LCT muffin was consumed within 15 min, and then 6-h meal tolerance test was conducted. The muffin had approximately 465 kcal, 8.36 g of protein, 17.24 g of fat, and 69.0 g of carbohydrate; among the 17.24g of fat, 15g of fat was LCT.
  Arms: LCT consumption
Dietary Supplement: MCDG oil — MCDG muffin was provided to the study participants. The MCDG muffin was consumed within 15 min, and then 6-h meal tolerance test was conducted. The muffin had approximately 465 kcal, 8.36 g of protein, 17.24 g of fat, and 69.0 g of carbohydrate; among the 17.24g of fat, 15g of fat was MCDG.
  Arms: MCDG consumption

SUMMARY:
It is well known that medium chain triglycerides (MCTs) and diacylglycerols (DGs) have effects on lowering circulating triglycerides (TGs). In this study, the mixture of MCTs and DGs (MCDGs) examined whether it has beneficial effects on postprandial lipids metabolism compared to long-chain triglycerides (TGs).

DETAILED DESCRIPTION:
A randomized, double-blinded, controlled, cross-over trial was conducted to verify the effects of MCDGs. Twenty-eight healthy male and female subjects aged 21-29 years with normal body weight [18.5 kg/m^2 ≤ body mass index (BMI) < 25 kg/m^2] were recruited. The subjects visited the research site twice over with a seven-day interval after an overnight fast at least 12 hr. On the first visit, the participants were randomly assigned to consume a test or placebo product [test product: muffins containing MCDG oil (MCDG muffin); placebo product: muffins containing LCT oil (LCT muffin)] and ingested the assigned product. On the second visit, the participants consumed the other product that they did not eat on the first visit. On both visit day, the 6-hr meal tolerance test was conducted and started at 8:00 in the morning; venous blood samples were collected before (0 hr) and after ingestion (2, 3, 4, and 6 hr) of the products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with normal body weight (18.5 kg/m^2 ≤ body mass index (BMI) < 25 kg/m^2)

Exclusion Criteria:

* history/presence of hypertension, diabetes mellitus, hyperlipidemia, cardiovascular disease, liver disease, gastrointestinal disease, thyroid disease, or any other acute or chronic diseases requiring treatment
* Use of any medication affecting body weight or energy expenditure for 1 month before screening

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Triglyceride levels | 6 hours
  Triglyceride level differences during the 6-hr meal tolerance test between LCT and MCDG muffins intake

SECONDARY OUTCOMES:
The areas under the curve (AUC) of triglycerides | 1 day of second visit (after finishing cross-over trial)
  Triglyceride AUC differences between LCT and MCDG muffins intake
Triglyceride maximum concentration time | 1 day of second visit (after finishing cross-over trial)
  The time when triglyceride peaks maximum concentration during the 6-h meal tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Jong Ho Lee, Ph.D, Principal Investigator — Yonsei University
Locations (1):
- Laboratory of Clinical Nutrigenetics/Nutrigenomics, Yonsei University., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No